CLINICAL TRIAL: NCT05231902
Title: Prevalence of Attention Deficit/Hyperactivity Disorder and Parenting Stress in School-age Children in Chongqing, China
Acronym: PADHDPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chen Li (Other)
Responsible Party: Sponsor-Investigator, Chen Li, Associate Professor，Director, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Other Study IDs: CHENl
Record Dates: First submitted 2022-01-30; First posted 2022-02-09 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: ADHD
Keywords: ADHD; parenting stress
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Attention deficit hyperactivity disorder (ADHD) is a common chronic neurodevelopmental disorder. Around 7.2% of children around the world are suffering from ADHD, while a chinese meta-analysis shows that the prevalence is 6.28%. There is no study of ADHD prevalence have used population-based samples, and depending on Vanderbilt ADHD Diagnostic Parent Rating Scale (VADPRS), in Chongqing, China. The purpose of the study is to investigate the prevalence of ADHD in school-age children and the parenting stress of parents of ADHD children in Chongqing. According to the proportion of primary school students in the four regions of Chongqing, using stratified proportional random sampling, 6480 primary school students are proposed to be selected as the research object, and questionnaires will complete by their caregivers and class teachers. VADPRS is used to evaluate the prevalence. Caregiver strain questionnaire (CGSQ) was used to assess parenting stress. Because of the nature of ADHD and the seriousness of its consequences, the periodic estimation of the prevalence of ADHD has been a critical research aim. This study can not only evaluate the prevalence of ADHD and parenting stress of parents of children with ADHD, but also use campus screening to promote parents and teachers' understanding of ADHD and improve the treatment rate.

DETAILED DESCRIPTION:
Background: Attention deficit hyperactivity disorder (ADHD) is a common chronic neurodevelopmental disorder in children. The global prevalence of ADHD in children and adolescents is about 7.2%, while a domestic meta-analysis shows that its prevalence is about 6.3%. Foreign studies have shown that the parenting stress of parents of ADHD children is significantly higher than that of normal children. Vanderbilt scale is developed according to DSM-IV ADHD diagnostic criteria and revised with the latest DSM-V. It is applicable to school-age children, including Vanderbilt ADHD diagnostic parent rating scale (VADPRS) and Vanderbilt ADHD diagnostic teachers rating scale (VADTRS). The previous single center study of our research group has verified the reliability and validity of Vanderbilt scale. At present, a domestic multi-center research is being carried out, and the scale has been used in the diagnosis of ADHD in many countries. The caregiver strain questionnaire (CGSQ) is applicable to assess the pressure of parents of children under the age of 18 due to their children's problems. The 21 items of CGSQ are divided into three dimensions to assess parenting pressure, including objective pressure, subjective internal pressure and subjective external pressure. Likert grade 5 score is adopted, with a total score of 21 ~ 105, The higher the score, the greater the parenting pressure of caregivers. Relevant studies have confirmed that the questionnaire can be used to evaluate the parenting pressure of parents of ADHD children. The children's sleep habits questionnaire (CSHQ) is compiled on the basis of referring to the international classification of sleep problems/disorders. It is applicable to the ages of 4 ~ 12 years. The 35 items of CSHQ (33 of which enter the scoring system) have 8 levels, reflecting the common sleep problems/disorders of children, which are filled in by the guardian according to the typical sleep performance of children in recent half a year, The total score of CSHQ ≥ 41 indicates that it is a sleep problem/disorder. One research showed that the measurement performance of CSHQ in the evaluation of sleep status of school-age children in China is relatively stable.

Objective and significance: To understand the positive rate and difference of VADPRS and VADTRS among school-age children in Chongqing; To understand the parenting stress of children with VADPRS positive. At present, domestic pay less attention to the parenting pressure of ADHD children's parents, and these parents have not received social support. The significance of this study is to kown the prevalence of ADHD in Chongqing, improve parents' and teachers' understanding of ADHD, finally improve the treatment rate of ADHD, and hope to give rise to more attention to the parenting pressure of parents of ADHD children in China.

Research design: The sample size of primary school students in Chongqing is randomly divided into four regions according to the proportion of each region. The parents' questionnaire includes basic information, VADPRS, CSHQ and CGSQ, and the teachers' questionnaire includes basic information and VADTRS.

Sample size calculation: the minimum sample size calculation formula is adopted N=μα2×π×（1-π）/δ2 The sample confirmation: According to the existing literature at home and abroad, the prevalence of ADHD in children and adolescents (π≈ 7%) is the basis for determining the sample size and allowable error(δ) = 0.15 π, α =0.05, μα=1.96 Sample size required: N=1.962×0.07×（1-0.07）/（0.07×0.15）2=2268 Assuming that the response rate is 70%, the expanded sample size is 3240. Because the stratified cluster random sampling method is adopted in this study, the sample size is doubled and 6480 people should be investigated.

Statistical analysis: All the data are analyzed using SPSS 26.0; The statistics adopt two-sided test, and the test level is 0.05. Continuous variables that conform to the normal distribution are described by mean ± standard deviation, those don't conform to the normal distribution are described by median (first and third quartiles), and the number of use cases (percentage) of classified variables are described; Paired t-test or Wilcoxon signed rank sum test were used for the comparison of paired data

Ethical matters and data protection: The parents and teachers of school-age students participated in the study will sign the informed consent. And this study was approved by the local ethics committee. Every participated student has a only code then the research data will be provided to the researcher. The authorization from parents on the patient's health information remains valid until the study is completed. After that, researchers will delete private information from the study record.

ELIGIBILITY:
Inclusion Criteria:

teacher: have been the teacher of the children more than one month; sign the informed consent

parent: children in the selected primary school; sign the informed consent

Exclusion Criteria:

parents: don't live with children

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: school-age student in the selected primary school
Sampling Method: Non-Probability Sample
Enrollment: 6480 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The positive rate of Vanderbilt ADHD Diagnostic Parent Rating Scale among school-age children in Chongqing | 6 months
  Vanderbilt ADHD diagnostic parent rating scale (VADPRS) includes two parts: behavior and performance. Behavior part: attention deficit (items 1 ~ 9), hyperactivity / impulse (items 10 ~ 18), are scored according to four levels of 0 ~ 3; The performance part includes 8 items, 4 items are used to evaluate the children's academic performance and 4 items are used to evaluate the children's interpersonal relationship, with a five grade score of 1 ~ 5 Attention deficit: from item 1 to 9, at least 6 items ≥ 2 score Hyperactivity impulse: from item 10 to 18, at least 6 items ≥ 2 score Functional impairment: at least 2 items ≥ 4 score or at least 1 item≥ 5 score Positive: meet attention deficit + functional impairment or hyperactivity impulse + functional impairment or attention deficit + hyperactivity/impulse+functional impairment
Parenting stress of parents of children with positive Vanderbilt ADHD Diagnostic Parent Rating Scale | 6 months
  The total score of 21 items in caregiver stress questionnaire (CGSQ) questionnaire is from 21 to 105, the higher total score, the greater the pressure. Compare the CGSQ score between VADPRS (+) and VADPRS (-).

SECONDARY OUTCOMES:
The positive rate of Vanderbilt ADHD diagnostic teacher rating scale for school-age children in Chongqing | 6 months
  Vanderbilt ADHD diagnostic teacher rating scale (VADTRS) includes two parts: behavior and performance. Behavior part: attention deficit (items 1 ~ 9), hyperactivity / impulse (items 10 ~ 18), are scored according to four levels of 0 ~ 3; The performance part includes 8 items, 4 items are used to evaluate the children's academic performance and 4 items are used to evaluate the children's interpersonal relationship, with a five grade score of 1 ~ 5 Attention deficit: from item 1 to 9, at least 6 items ≥ 2 score Hyperactivity impulse: from item 10 to 18, at least 6 items ≥ 2 score Functional impairment: at least 2 items ≥ 4 score or at least 1 item≥ 5 score Positive: meet attention deficit + functional impairment or hyperactivity impulse + functional impairment or attention deficit + hyperactivity/impulse+functional impairment
Sleep status of children with Vanderbilt ADHD diagnostic parent rating scale positive screening | 6 months
  The total score is the sum of the scores of 33 items of child sleep habit questionnaire (CSHQ). If the total score is ≥ 41, it is positive. VADPRS (+) and VADPRS (-) compare the positive situation of CSHQ
Parenting stress of children with both positive Vanderbilt ADHD diagnostic parent rating scale and positive child sleep habit questionnaire | 6 months
  In Vanderbilt ADHD diagnostic parent rating scale (VADPRS) (+), compare caregiver stress questionnaire(CGSQ) score between child sleep habit questionnaire (CSHQ) (+) and child sleep habit questionnaire (CSHQ) (-). The higher score, the greater stress.

CONTACTS AND LOCATIONS:
Overall Officials: Li Chen, doctor, Study Director — Children's Hospital of Chongqing Medical University
Locations (1):
- Growth, Development and Mental health of Children and Adolescence Center, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data is confidential during the study

REFERENCES:
- [Background] Wolraich ML, Hagan JF Jr, Allan C, Chan E, Davison D, Earls M, Evans SW, Flinn SK, Froehlich T, Frost J, Holbrook JR, Lehmann CU, Lessin HR, Okechukwu K, Pierce KL, Winner JD, Zurhellen W; SUBCOMMITTEE ON CHILDREN AND ADOLESCENTS WITH ATTENTION-DEFICIT/HYPERACTIVE DISORDER. Clinical Practice Guideline for the Diagnosis, Evaluation, and Treatment of Attention-Deficit/Hyperactivity Disorder in Children and Adolescents. Pediatrics. 2019 Oct;144(4):e20192528. doi: 10.1542/peds.2019-2528. PMID 31570648
- [Background] Liu A, Xu Y, Yan Q, Tong L. The Prevalence of Attention Deficit/Hyperactivity Disorder among Chinese Children and Adolescents. Sci Rep. 2018 Aug 16;8(1):11169. doi: 10.1038/s41598-018-29488-2. PMID 30115972
- [Background] Leitch S, Sciberras E, Post B, Gerner B, Rinehart N, Nicholson JM, Evans S. Experience of stress in parents of children with ADHD: A qualitative study. Int J Qual Stud Health Well-being. 2019 Dec;14(1):1690091. doi: 10.1080/17482631.2019.1690091. PMID 31713473
- [Background] Bussing R, Gary FA, Mason DM, Leon CE, Sinha K, Garvan CW. Child temperament, ADHD, and caregiver strain: exploring relationships in an epidemiological sample. J Am Acad Child Adolesc Psychiatry. 2003 Feb;42(2):184-92. doi: 10.1097/00004583-200302000-00012. PMID 12544178
- [Background] Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000 Dec 15;23(8):1043-51. PMID 11145319
- [Derived] Tan J, Yi W, Shen J, Peng B, Gong M, Li F, Chen L. Impact of online health education on attention-deficit/hyperactivity disorder screening results and parenting stress among school-aged children. Front Psychiatry. 2025 Jan 31;16:1522263. doi: 10.3389/fpsyt.2025.1522263. eCollection 2025. PMID 39958151